CLINICAL TRIAL: NCT00413478
Title: Phase II Study of 5-Azacytidine (Azacytidine; Vidaza) in Chronic Lymphocytic Leukemia
Brief Title: 5-Azacytidine (Azacytidine; Vidaza) in Chronic Lymphocytic Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0428; NCI-2010-00552 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2006-12-15; First posted 2006-12-19 (Estimated); Results first posted 2015-06-30 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Chronic Lymphocytic Leukemia; Leukemia
Keywords: 5-Aza; Azacytidine; Vidaza; CLL; Chronic Lymphocytic Leukemia; Richter's transformation; Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 5-Azacytidine (Experimental): 5-Azacytidine 75mg/m^2 subcutaneously daily for seven days. Treatment cycles will be repeated every 3-8 weeks.
  Interventions: Drug: 5-Azacytidine

INTERVENTIONS:
Drug: 5-Azacytidine — Starting dose level: 75mg/m^2 subcutaneously daily for seven days. Treatment cycles will be repeated every 3-8 weeks.
  Other Names: Azacytidine; Vidaza; 5-aza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816

SUMMARY:
The objective of this study is to determine the safety and efficacy of Azacytidine in fludarabine-resistant chronic lymphocytic leukemia (CLL), Richter's transformation, and T-cell prolymphocytic leukemia (T-PLL).

DETAILED DESCRIPTION:
Azacytidine is designed to block certain genes in cancer cells whose job is to stop the function of the tumor-fighting genes. By blocking the "bad" genes, the tumor-fighting genes may be able to work better.

Before you can start treatment on this study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. You will have blood drawn (about 3 teaspoons) to check your kidney and liver function (routine blood tests). You may have a bone marrow aspiration performed (if you have not had one in recent weeks). To collect a bone marrow aspirate, an area of the hip or chest bone is numbed with anesthetic, and a small amount of bone marrow is withdrawn through a large needle. Women who are able to have children must have a negative urine pregnancy test.

If you agree to take part in this study, you will receive azacytidine by subcutaneous (just under the skin) injection every day for 7 days. This course of treatment will be repeated every 3-8 weeks, depending on the results of your routine blood tests.

Your doctor may increase or decrease your dose of azacytidine, depending on if you experience any side effects. You will continue to receive treatment on this study unless the disease gets worse or you experience any intolerable side effects. If the disease gets worse or you experience any intolerable side effects, you will be taken off this study.

This is an investigational study. This is an investigational study. Azacytidine has been approved by the FDA for the treatment of myelodysplastic syndrome. Up to 37 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic lymphocytic leukemia (CLL), prolymphocytic leukemia, Richter's transformation or T-PLL who have previously been treated with fludarabine or another regime are eligible.
2. Patients with histologically or cytologically confirmed Richter's transformation.
3. Serum glutamic-oxaloacetic transaminase (SGOT) or serum glutamic-pyruvic transaminase (SGPT) less than x 2 normal levels.
4. Women of childbearing potential who have a negative pregnancy test prior to azacytidine treatment.
5. Women of childbearing potential who agreed not to become pregnant and men agreed not to father a child while on azacytidine treatment.
6. Performance 0-2 (ECOG). Adequate liver function (bilirubin of less than2mg/dl) and renal function (creatinine less than 2mg/dl). Adequate cardiac functions (NYHA cardiac III-IV excluded).
7. Signed informed consent.

Exclusion Criteria:

1. Breast feeding or pregnant females. Patients of (male and female) childbearing potential should practice effective methods of contraception; otherwise, they will be excluded. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
2. Known or suspected hypersensitivity to azacytidine or Mannitol.
3. Active and uncontrolled infections.
4. Patients with advanced malignant hepatic tumors.
5. Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zeev Estrov, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Malik A, Shoukier M, Garcia-Manero G, Wierda W, Cortes J, Bickel S, Keating MJ, Estrov Z. Azacitidine in fludarabine-refractory chronic lymphocytic leukemia: a phase II study. Clin Lymphoma Myeloma Leuk. 2013 Jun;13(3):292-5. doi: 10.1016/j.clml.2012.11.009. Epub 2012 Dec 21. PMID 23265768
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 09/21/2006 to 12/01/2010. All recruitment done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: The study was discontinued after 9 participants enrolled because of lack of efficacy and slow accrual.
Groups:
- 5-Azacytidine: 5-Azacytidine 75 mg/m^2 subcutaneously daily for 7 days, cycle repeated every 3-8 weeks.
Period: Overall Study
Arm/Group | 5-Azacytidine
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 5-Azacytidine
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: years] | 74 [49 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response Rate (Complete, Partial) of Azacytidine
Description: Overall response rate includes percentage of participants with complete response (CR) plus partial response (PR) responses using the National Cancer Institute (NCI) International Workshop on Chronic Lymphocytic Leukemia (IWCLL) criteria for response: Complete response defined as no palpable lymph nodes, liver or spleen and absence of symptoms. Neutrophil count > 15,00/Mic L, and platelet count more than 100,000/MicL. Hemoglobin should be > 11g/dl without transfusions. Lymphocyte count <4000/micL. On bone marrow aspirate lymphocyte % should be <30%, and biopsy showing no lymphocyte infiltrate. A partial response was defined as more than or equal to 50% decrease in lymph nodes and liver and spleen size. Neutrophils > 1500/ micL or >50 % improvement from baseline, platelet count >100,000/micL or >50 % improvement from baseline. Hemoglobin >11g/dl or >50% improvement from baseline. A reduction of >50% in Leukocyte count or <30 % lymphocytes with residual disease on biopsy for nodular PR.
Time Frame: 3 to 8 weeks treatment cycles, continuation up to 1 year
Measure: Number; unit: percentage of participants
Arm/Group | 5-Azacytidine
Number analyzed (Participants) | 9
percentage of participants | 0

ADVERSE EVENTS:
Time Frame: Adverse event data collected with each 7 day treatment through subsequent repeated treatment cycles every 3 to 8 weeks with continuation up to 1 year. Overall collection period: October 2006 to August 2009.
Arm/Group | 5-Azacytidine
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 9/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 5-Azacytidine (N=9)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 3
Diarrhea (Gastrointestinal disorders) | 2
Skin Rash (Skin and subcutaneous tissue disorders) | 3
Infections (Infections and infestations) | 6
Fever (General disorders) | 2
Pneumonia (Infections and infestations) | 3
Vomiting (Gastrointestinal disorders) | 2
Arrythmia (Cardiac disorders) | 1
Bells Palsy (Nervous system disorders) | 1
blurry vision (Eye disorders) | 1
Cellulitis (Infections and infestations) | 1
Constipation (Gastrointestinal disorders) | 1
cramps (Musculoskeletal and connective tissue disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
dysuria (Renal and urinary disorders) | 1
Edema (Vascular disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
fatigue (General disorders) | 1
headache (General disorders) | 1
Hematoma (Blood and lymphatic system disorders) | 1
Hypomagnesia (Metabolism and nutrition disorders) | 1
lightheadedness (General disorders) | 1
MRSA Infection (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 3
Neutropenic fever (Infections and infestations) | 1
Pain (General disorders) | 1
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Infiltrates (Infections and infestations) | 1
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 3
Sweats (General disorders) | 1
swollen lips (General disorders) | 1
weight loss (Gastrointestinal disorders) | 1

LIMITATIONS AND CAVEATS:
Early termination led to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes